CLINICAL TRIAL: NCT01569568
Title: Investigation of Brain Nitrogen in Partial Ornithine Transcarbamylase Deficiency (OTCD) Using 1 H MRS, DTI, and fMRI
Status: Completed | Type: Observational
Sponsor: Andrea Gropman (Other)
Collaborators: Children's National Research Institute (Other)
Responsible Party: Sponsor-Investigator, Andrea Gropman, MD, Children's National Research Institute
Organization: Children's National Research Institute (Other)
Other Study IDs: UCRDC 5107
Record Dates: First submitted 2012-03-30; First posted 2012-04-03 (Estimated); Results first posted 2017-04-14 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-02

CONDITIONS: Ornithine Transcarbamylase Deficiency
Keywords: Neuroimaging; MRI; Urea cycle; hyperammonemia; cognitive function; ornithine transcarbamylase deficiency
MeSH Terms: conditions — Ornithine Carbamoyltransferase Deficiency Disease; Hyperammonemia | interventions — Neuropsychological Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Subjects with OTCD: males and females ages 7-60 years with OTCD who are able to undergo MRI and cognitive testing MRI scanning
  1H MRS, DTI, FMRI Cognitive testing Neuropsychological testing
  Interventions: Other: MRI scanning; Behavioral: Cognitive testing
- Healthy controls: males and females ages 7-60 years who are healthy controls who are able to undergo MRI and cognitive testing MRI scanning
  1H MRS, DTI, FMRI Cognitive testing Neuropsychological testing
  Interventions: Other: MRI scanning; Behavioral: Cognitive testing

INTERVENTIONS:
Other: MRI scanning — 1H MRS, DTI, FMRI
  Other Names: MRI
Behavioral: Cognitive testing — Behavioral testing

SUMMARY:
The purpose of this study is to use various types of MRI and cognitive testing to evaluate changes in the brain and cognitive function that occur in subjects with ornithine transcarbamylase deficiency (OTCD) relative to healthy individuals

DETAILED DESCRIPTION:
The overall goal of this project is to characterize metabolic, structural and cognitive changes in OTCD using 1H MRS, DTI, volumetric averaging and fMRI with cognitive testing of executive function measures to validate biomarkers for the effect of HA and its treatment on the brain.

The investigators will measure gln and mI in blood and brain (using 1H MRS) in affected participants, and mI in brain in controls, fractional anisotropy as a measure of white matter microstructural damage (by DTI) and brain activation pathways alterations with tasks probing working memory (fMRI). As a secondary outcome measure, the investigators will correlate the findings from neuroimaging with cognitive functioning. This protocol is based on the previous 5104 protocol, now includes children to evaluate the age and stage of disease on these indices in a cohort that is undergoing important developmental events against an age matched typically developing cohort.

ELIGIBILITY:
Inclusion Criteria:

Subject inclusion criteria:

1. Patients with OTCD;
2. Age range: 7-60 years
3. Able to undergo neuroimaging safely (i.e. without presence of ferromagnetic devices)
4. Subject has a documented full scale IQ > 70

Control participant inclusion criteria:

1. Healthy males and females without metabolic disease aged 7-60 years
2. Subject has a documented full scale IQ > 70

Exclusion Criteria:

Subject exclusion criteria:

1. Mental retardation (i.e., Full Scale IQ< 70)
2. Age range <7 or >60 years
3. Presence of ferromagnetic device(s) that preclude safe imaging
4. Pregnant female

Control exclusion criteria:

1. Subjects with a documented history of an intellectual deficit (i.e., Full Scale IQ< 70)
2. Age range <7 or >60 years
3. Presence of ferromagnetic device(s) that preclude safe imaging
4. Pregnant female

Ages: 7 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Males and females, ages 7-60 years with ornithine transcarbamylase deficiency Males and females, ages 7-60 years who are healthy controls without ornithine transcarbamylase deficiency
Sampling Method: Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2010-09; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea L Gropman, M.D., Principal Investigator — Children's National Research Institute

IPD SHARING:
Plan to Share IPD: Yes
Final data is on the UCDC website

REFERENCES:
- [Background] Gropman AL, Shattuck K, Prust MJ, Seltzer RR, Breeden AL, Hailu A, Rigas A, Hussain R, VanMeter J. Altered neural activation in ornithine transcarbamylase deficiency during executive cognition: an fMRI study. Hum Brain Mapp. 2013 Apr;34(4):753-61. doi: 10.1002/hbm.21470. Epub 2011 Nov 23. PMID 22110002
- [Background] Prust MJ, Gropman AL, Hauser N. New frontiers in neuroimaging applications to inborn errors of metabolism. Mol Genet Metab. 2011 Nov;104(3):195-205. doi: 10.1016/j.ymgme.2011.06.020. Epub 2011 Jun 30. PMID 21778100
- [Background] Gropman AL, Gertz B, Shattuck K, Kahn IL, Seltzer R, Krivitsky L, Van Meter J. Diffusion tensor imaging detects areas of abnormal white matter microstructure in patients with partial ornithine transcarbamylase deficiency. AJNR Am J Neuroradiol. 2010 Oct;31(9):1719-23. doi: 10.3174/ajnr.A2122. Epub 2010 May 20. PMID 20488904
- [Background] Gropman A. Brain imaging in urea cycle disorders. Mol Genet Metab. 2010;100 Suppl 1(Suppl 1):S20-30. doi: 10.1016/j.ymgme.2010.01.017. Epub 2010 Feb 13. PMID 20207564
- [Background] Oldham MS, VanMeter JW, Shattuck KF, Cederbaum SD, Gropman AL. Diffusion tensor imaging in arginase deficiency reveals damage to corticospinal tracts. Pediatr Neurol. 2010 Jan;42(1):49-52. doi: 10.1016/j.pediatrneurol.2009.07.017. PMID 20004862
- [Background] Gropman AL, Sailasuta N, Harris KC, Abulseoud O, Ross BD. Ornithine transcarbamylase deficiency with persistent abnormality in cerebral glutamate metabolism in adults. Radiology. 2009 Sep;252(3):833-41. doi: 10.1148/radiol.2523081878. Epub 2009 Jun 30. PMID 19567648
- [Background] Gropman AL, Fricke ST, Seltzer RR, Hailu A, Adeyemo A, Sawyer A, van Meter J, Gaillard WD, McCarter R, Tuchman M, Batshaw M; Urea Cycle Disorders Consortium. 1H MRS identifies symptomatic and asymptomatic subjects with partial ornithine transcarbamylase deficiency. Mol Genet Metab. 2008 Sep-Oct;95(1-2):21-30. doi: 10.1016/j.ymgme.2008.06.003. Epub 2008 Jul 26. PMID 18662894
- See also: Family support group — http://NUCDF.org
- See also: Urea Cycle rare disease consortium — https://ucdc.rarediseasesnetwork.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Subjects With OTCD: males and females ages 7-60 years with OTCD
  MRI scanning: 1H Magnetic Resonance Spectroscopy (MRS), Diffusion Tensor Imaging (DTI), functional magnetic resonance imaging (fMRI)
  Cognitive testing: Neuropsychological testing
- Healthy Controls: males and females ages 7-60 years who are healthy controls
  MRI scanning: 1H MRS, DTI, FMRI
  Cognitive testing: Neuropsychological testing
Period: Overall Study
Arm/Group | Subjects With OTCD | Healthy Controls
Started | 20 | 29
Completed | 20 | 27
Not Completed | 0 | 2
Not completed — Physician Decision | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Subjects With OTCD: males and females ages 7-60 years with OTCD
  MRI scanning: 1H MRS, DTI, FMRI
  Cognitive testing: Neuropsychological testing
- Total: Total of all reporting groups
Arm/Group | Subjects With OTCD | Healthy Controls | Total
Number analyzed (Participants) | 20 | 27 | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.3 (19.4) | 25.8 (14.6) | 28.05 (17.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 19 | 36
  Male | 3 | 8 | 11

OUTCOME MEASURES:

1. Primary Outcome: Concentration of Glutamine and Myoinositol
Description: Concentration based on area under curve on 1H Magnetic Resonance Spectroscopy(MRS) and quantitated by LCModel (a method that allows automatic quantitation of spectroscopy data). A metabolite's tissue concentration is related to the integrated amplitude, the area under the curve of the MRS signal, it produces. While MRS signals are usually acquired in the time domain as free induction decays or echoes, they are usually viewed and analyzed in the frequency domain. The frequency domain representation is derived from the acquired time domain data by the Fourier Transform. The protocol we use selects 257 averages. The machine summates the data at each time point to generate one value for the area under the curve. Therefore, we don't have the measurement at each time point.
  Furthermore, we measured voxels in two different brain areas containing different kinds of brain matter: one voxel was located in posterior cingulate gray matter (PCGM) and the other in parietal white matter (PWM).
Time Frame: Baseline
Population: Two OTCD patients and one healthy control were excluded due to excessive head motion.
Measure: Mean (Standard Deviation); unit: mM
Arm/Group | Subjects With OTCD | Healthy Controls
Number analyzed (Participants) | 18 | 26
mM
  Concentration of glutamine in PWM | 2.61 (1.07) | 1.66 (0.93)
  Concentration of myoinositol in PWM | 2.23 (0.84) | 2.69 (0.48)
  Concentration of glutamine in PCGM | 5.22 (1.70) | 3.62 (0.91)
  Concentration of myoinositol in PCGM | 3.80 (0.80) | 4.37 (0.46)
Statistical Analysis 1: Comparison: Subjects With OTCD vs Healthy Controls; The null hypothesis predicts that the concentration of glutamine is the same for controls and OTCD patients in PCGM; Test type: Superiority or Other; p = 0.001, t-test, 2 sided — This is an uncorrected p-value. A priori threshold is 0.05
Statistical Analysis 2: Comparison: Subjects With OTCD vs Healthy Controls; The null hypothesis predicts that the concentration of myoinositol is the same for controls and OTCD patients in PCGM; Test type: Superiority or Other; p = 0.011, t-test, 2 sided — This is an uncorrected p-value. A priori significance threshold is 0.05
Statistical Analysis 3: Comparison: Subjects With OTCD vs Healthy Controls; The null hypothesis predicts that the concentration of glutamine is the same for controls and OTCD patients in PWM; Test type: Superiority or Other; p = 0.004, t-test, 2 sided — This is an uncorrected p-value. A priori threshold was 0.05
Statistical Analysis 4: Comparison: Subjects With OTCD vs Healthy Controls; The null hypothesis predicts that the concentration of myoinositol is the same for controls and OTCD patients in PWM; Test type: Superiority or Other; p = 0.046, t-test, 2 sided — This is an uncorrected p-value. A priori threshold was 0.05

2. Primary Outcome: Functional Connectivity of Assessed by Resting-state fMRI
Description: Investigation of differences in functional connectivity of OTCD patients compared to healthy controls, particularly in the default-mode network (DMN) and the set-maintenance network (SMN). Participants underwent a resting-state scan using 3T fMRI. Combining independent component analysis (ICA) and region-of-interest (ROI) analyses, identified the nodes that comprised each network in each group, and assessed internodal connectivity. For each subject, this analysis generated a correlation value, which reflected the strength of functional connectivity between each ROI pair.The correlation r-values were normalized using Fisher's r-to-Z-transform, generating z-scores. The DMN was composed of 1) anterior cingulate/medial prefrontal cortex (ACC/mPFC), 2) posterior cingulate cortex (PCC), and 3) bilateral inferior parietal lobule (IPL). The SMN was composed of 1)ACC, 2) bilateral superior frontal gyrus (SFG), and 3) bilateral anterior insula/frontal operculum (aI/fO).
Time Frame: Baseline
Population: Resting state data was not acquired for several of our participants (7 controls and 4 patients). Furthermore, 3 OTCD patients were excluded from the analyses due to excessive head motion.
Measure: Mean (Standard Deviation); unit: z-scores
Arm/Group | Subjects With OTCD | Healthy Controls
Number analyzed (Participants) | 13 | 22
z-scores
  DMN: ACC/mPFC & left IPL connectivity | -0.86 (0.70) | 0.18 (0.30)
  DMN: ACC/mPFC & PCC connectivity | -0.10 (0.70) | 0.12 (0.40)
  DMN: ACC/mPFC & right IPL connectivity | -0.26 (0.53) | 0.07 (0.34)
  DMN: PCC & left IPL connectivity | 0.69 (0.63) | 0.69 (0.31)
  DMN: PCC & right IPL connectivity | 0.66 (0.42) | 0.64 (0.30)
  DMN: left IPL & right IPL connectivity | 0.75 (0.69) | 0.70 (0.34)
  SMN: ACC & left aI/fO connectivity | 0.19 (0.39) | 0.28 (0.41)
  SMN: ACC & left SFG connectivity | 0.28 (0.35) | 0.44 (0.29)
  SMN: ACC & right aI/fO connectivity | 0.21 (0.30) | 0.44 (0.29)
  SMN: ACC & right SFG connectivity | 0.29 (0.37) | 0.59 (0.23)
  SMN: left aI/fO & left SFG connectivity | 0.10 (0.35) | 0.22 (0.38)
  SMN: left aI/fO & right aI/fO connectivity | 0.71 (0.43) | 0.80 (0.35)
  SMN: left aI/fO & right SFG connectivity | 0.05 (0.33) | 0.11 (0.33)
  SMN: left SFG & right SFG connectivity | 0.70 (0.43) | 0.68 (0.28)
  SMN: right aI/fO & left SFG connectivity | 0.02 (0.22) | 0.25 (0.21)
  SMN: right aI/fO & right SFG connectivity | 0.04 (0.26) | 0.27 (0.35)
Statistical Analysis 1: Comparison: Subjects With OTCD vs Healthy Controls; The null hypothesis states predicts no main effects of Group, ROI pair, or Age, suggesting that the connectivity between all DMN nodes is the same across groups; Test type: Superiority or Other; p < 0.001, ANOVA — Our a priori threshold for statistical significance was 0.05; We ran a 2 (Group) x 6 (ROI Pair) ANOVA to assess functional connectivity between the nodes of the DMN, using age as a covariate
Statistical Analysis 2: Comparison: Subjects With OTCD vs Healthy Controls; The null hypothesis predicts that functional connectivity between the ACC/mPFC node and the left IPL node does not differ between groups; Test type: Superiority or Other; p = 0.024, ANOVA — This is an uncorrected p-value. A priori significance threshold was 0.05; We ran a series of post-hoc one-way ANOVAs to localize the main effect found. Age was used as a covariate
Statistical Analysis 3: Comparison: Subjects With OTCD vs Healthy Controls; The null hypothesis predicts that functional connectivity between the ACC/mPFC node and the PCC node does not differ between groups; Test type: Superiority or Other; p = 0.040, ANOVA — This is an uncorrected p-value. A priori significance threshold is 0.05; We ran a series of post-hoc one-way ANOVAs to localize the main effect found. Age was used as a covariate
Statistical Analysis 4: Comparison: Subjects With OTCD vs Healthy Controls; The null hypothesis predicts that functional connectivity between the ACC/mPFC node and the right IPL node does not differ between groups; Test type: Superiority or Other; p = 0.008, ANOVA — This is an uncorrected p-value. A priori significance threshold was 0.05; We ran a series of post-hoc one-way ANOVAs to localize the main effect found. Age was used as a covariate
Statistical Analysis 5: Comparison: Subjects With OTCD vs Healthy Controls; The null hypothesis predicts that functional connectivity between the left IPL node and the right IPL node does not differ between groups; Test type: Superiority or Other; p = 0.470, ANOVA — This is an uncorrected p-value. A priori significance threshold was 0.05; We ran a series of post-hoc one-way ANOVAs to localize the main effect found. Age was used as a covariate
Statistical Analysis 6: Comparison: Subjects With OTCD vs Healthy Controls; The null hypothesis predicts that functional connectivity between the PCC node and the left IPL node does not differ between groups; Test type: Superiority or Other; p = 0.829, ANOVA — This is an uncorrected p-value. A priori significance threshold was 0.05; We ran a series of post-hoc one-way ANOVAs to localize the main effect found. Age was used as a covariate
Statistical Analysis 7: Comparison: Subjects With OTCD vs Healthy Controls; The null hypothesis predicts that functional connectivity between the PCC node and the right IPL node does not differ between groups; Test type: Superiority or Other; p = 0.801, ANOVA — This is an uncorrected p-value. A priori significance threshold was 0.05; We ran a series of post-hoc one-way ANOVAs to localize the main effect found. Age was used as a covariate
Statistical Analysis 8: Comparison: Subjects With OTCD vs Healthy Controls; The null hypothesis states predicts no main effects of Group, ROI pair, or Age, suggesting that the connectivity between all SMN nodes is the same across groups; Test type: Superiority or Other; p < 0.001, ANOVA — Our a priori threshold for statistical significance was 0.05; We ran a 2 (Group) x 6 (ROI Pair) ANOVA to assess functional connectivity between the nodes of the SMN, using age as a covariate
Statistical Analysis 9: Comparison: Subjects With OTCD vs Healthy Controls; The null hypothesis predicts that functional connectivity between the ACC node and the left aI/fO node does not differ between groups; Test type: Superiority or Other; p = 0.550, ANOVA — This is an uncorrected p-value. A priori significance threshold was 0.05; We ran a series of post-hoc one-way ANOVAs to localize the main effect found. Age was used as a covariate
Statistical Analysis 10: Comparison: Subjects With OTCD vs Healthy Controls; The null hypothesis predicts that functional connectivity between the ACC node and the left SFG node does not differ between groups; Test type: Superiority or Other; p = 0.113, ANOVA — This is an uncorrected p-value. A priori significance threshold was 0.05; We ran a series of post-hoc one-way ANOVAs to localize the main effect found. Age was used as a covariate
Statistical Analysis 11: Comparison: Subjects With OTCD vs Healthy Controls; The null hypothesis predicts that functional connectivity between the ACC node and the right aI/fO node does not differ between groups; Test type: Superiority or Other; p = 0.039, ANOVA — This is an uncorrected p-value. A priori significance threshold was 0.05; We ran a series of post-hoc one-way ANOVAs to localize the main effect found. Age was used as a covariate
Statistical Analysis 12: Comparison: Subjects With OTCD vs Healthy Controls; The null hypothesis predicts that functional connectivity between the ACC node and the right SFG node does not differ between groups; Test type: Superiority or Other; p = 0.005, ANOVA — This is an uncorrected p-value. A priori significance threshold was 0.05; We ran a series of post-hoc one-way ANOVAs to localize the main effect found. Age was used as a covariate
Statistical Analysis 13: Comparison: Subjects With OTCD vs Healthy Controls; The null hypothesis predicts that functional connectivity between the left aI/fO and the left SFG node does not differ between groups; Test type: Superiority or Other; p = 0.426, ANOVA — This is an uncorrected p-value. A priori significance threshold was 0.05; We ran a series of post-hoc one-way ANOVAs to localize the main effect found. Age was used as a covariate
Statistical Analysis 14: Comparison: Subjects With OTCD vs Healthy Controls; The null hypothesis predicts that functional connectivity between the left aI/fO node and the right aI/fO node does not differ between groups; Test type: Superiority or Other; p = 0.256, ANOVA — This is an uncorrected p-value. A priori significance threshold was 0.05; We ran a series of post-hoc one-way ANOVAs to localize the main effect found. Age was used as a covariate
Statistical Analysis 15: Comparison: Subjects With OTCD vs Healthy Controls; The null hypothesis predicts that functional connectivity between the left aI/fO and the right SFG node does not differ between groups; Test type: Superiority or Other; p = 0.853, ANOVA — This is an uncorrected p-value. A priori significance threshold was 0.05; We ran a series of post-hoc one-way ANOVAs to localize the main effect found. Age was used as a covariate
Statistical Analysis 16: Comparison: Subjects With OTCD vs Healthy Controls; The null hypothesis predicts that functional connectivity between the right aI/fO node and the left SFG node does not differ between groups; Test type: Superiority or Other; p = 0.003, ANOVA — This is an uncorrected p-value. A priori significance threshold was 0.05; We ran a series of post-hoc one-way ANOVAs to localize the main effect found. Age was used as a covariate
Statistical Analysis 17: Comparison: Subjects With OTCD vs Healthy Controls; The null hypothesis predicts that functional connectivity between the right aI/fO node and the right SFG node does not differ between groups; Test type: Superiority or Other; p = 0.023, ANOVA — This is an uncorrected p-value. A priori significance threshold was 0.05; We ran a series of post-hoc one-way ANOVAs to localize the main effect found. Age was used as a covariate

3. Primary Outcome: Fractional Anisotropy Assessed Using DTI
Description: Fractional Anisotropy (FA) is a measure of the diffusion asymmetry within a voxel as defined by its eigenvalues. In our study, FA is being used as a measure of white matter integrity, because FA is very sensitive to small microstructural changes.Fractional anisotropy (FA) is a scalar value between zero and one (0-1) that describe anisotropy of a diffusion process. A value of zero means that diffusion is isotropic, i.e. it is unrestricted (or equally restricted) in all directions. A value of one means that diffusion occurs only along one axis and is fully restricted along all other directions.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Subjects With OTCD | Healthy Controls
Number analyzed (Participants) | 20 | 27
units on a scale | 0.25 (0.003) | 0.3 (0.008)

4. Secondary Outcome: Neuropsychological Assessment
Description: Testing consisted of the Wechsler Abbreviated Scale of Intelligence (WASI), Comprehensive Trail Making Test (CTMT) (range 17-87), and the Behavioral Rating Inventory of Executive Function (BRIEF) (range GEC: 70-210; BRI:39-82 ; MI:41-92). The WASI includes three measures of intelligence; including, performance IQ (sum of block design and matrices sub scales; range: 40-160), verbal IQ (sum of vocabulary and similarities sub scales; range 40-160), and total IQ (sum of all four subscales; range: 80-320). The CTMT measures simple attention and executive function, it consists of five dot to dots that increase with complexity and difficulty. Higher values indicate better outcomes for all scales.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Subjects With OTCD | Healthy Controls
Number analyzed (Participants) | 20 | 29
units on a scale
  WASI - Verbal IQ | 107.33 (14.52) | 107.77 (18.59)
  WASI - Performance IQ | 98.5 (13.14) | 112.59 (14.54)
  WASI - Full IQ | 103.28 (14.02) | 111.22 (16.89)
  Trails - Composite | 48 (15) | 47 (12)
  Brief - Behavioral Regulation Index (BRI) | 55.59 (9.49) | 46.73 (8.90)
  Brief - Metacognition Index (MI) | 60.45 (11.75) | 47.38 (8.22)
  Brief - Global Executive Composite Score (GEC) | 59.05 (10.37) | 46.88 (7.67)
Statistical Analysis 1: Comparison: Subjects With OTCD vs Healthy Controls; Test type: Superiority or Other; p = .929, t-test, 2 sided — Equal variance is not assumed. Two tailed t-test WASI verbal IQ between cases and controls
Statistical Analysis 2: Comparison: Subjects With OTCD vs Healthy Controls; Test type: Superiority or Other; p = .002, t-test, 2 sided — Equal variance not assumed. Comparison WASI performance IQ cases and controls
Statistical Analysis 3: Comparison: Subjects With OTCD vs Healthy Controls; Test type: Superiority or Other; p = .094, t-test, 2 sided — Equal variance not assumed. Comparison of WASI full IQ cases and controls
Statistical Analysis 4: Comparison: Subjects With OTCD vs Healthy Controls; Test type: Superiority or Other; p = .853, t-test, 2 sided — Equal variance not assumed. Comparison of CTMT global composite score between cases and controls
Statistical Analysis 5: Comparison: Subjects With OTCD vs Healthy Controls; Test type: Superiority or Other; p = .001, t-test, 2 sided — Equal variance not assumed. Comparison of BRIEF BRI cases and controls
Statistical Analysis 6: Comparison: Subjects With OTCD vs Healthy Controls; Test type: Superiority or Other; p < .001, t-test, 2 sided — Equal variances not assumed. Comparison of BRIEF MI cases and controls
Statistical Analysis 7: Comparison: Subjects With OTCD vs Healthy Controls; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — Equal variances not assumed. Comparison of BRIEF GEC between cases and controls

ADVERSE EVENTS:
Arm/Group | Subjects With OTCD | Healthy Controls
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/29
Other Adverse Events (participants affected / at risk) | 0/20 | 0/29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No